CLINICAL TRIAL: NCT06363357
Title: The Effect of a Muscle-mimicking, Fabric-type Shoulder Orthosis on Functional Movements of the Upper Limb in Patients With Neuromuscular Disorder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Woo Hyung Lee, Assistant professor (MD, PhD), Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 24B-007-0000
Record Dates: First submitted 2024-04-09; First posted 2024-04-12 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-07

CONDITIONS: Muscular Dystrophy, Duchenne; Orthotic Devices; Upper Extremity; Neuromuscular Diseases (NMD); Fascioscapulohumeral Muscular Dystrophy; Spinal Muscular Atrophy (SMA); ALS (Amyotrophic Lateral Sclerosis); LGMD; SCI - Spinal Cord Injury
MeSH Terms: conditions — Muscular Dystrophy, Duchenne; Neuromuscular Diseases; Muscular Dystrophy, Facioscapulohumeral; Muscular Atrophy, Spinal; Amyotrophic Lateral Sclerosis; Spinal Cord Injuries

STUDY DESIGN:
Intervention Model Description: This study compares variables before and after wearing the shoulder orthosis in patients with neuromuscular disorder.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neuromuscular disorder participants (Experimental): This study compares variables before and after wearing the shoulder orthosis in patients with neuromuscular disorder.
  Interventions: Device: Shoulder orthosis

INTERVENTIONS:
Device: Shoulder orthosis — muscle-mimicking, fabric-type shoulder orthosis

SUMMARY:
The goal of this clinical trial is to investigate the effect of a muscle-mimicking, fabric-type shoulder orthosis on functional movements of the upper limb in patients with neuromuscular disorder.

The main questions it aims to answer are:

* What is the impact of the muscle-mimicking, fabric-type shoulder orthosis on upper limb functional movements in patients with neuromuscular disorder?
* Are there observable differences in upper limb function when the shoulder orthosis is worn versus when it is not?

Participants will:

* Receive education on how to wear and use the shoulder orthosis.
* Undergo evaluations, including assessment of upper limb performance, shoulder muscle strength testing, active range of motion measurements, assessment of functional workspace, goal attainment scale evaluation, surface electromyography, physiological measurements such as blood pressure and heart rate, fatigue assessment, and assessment for any musculoskeletal or skin-related issues.

Researchers will compare neuromuscular disorder patients before and while wearing and operating the shoulder orthosis to see if there are any significant effects on variables such as upper limb function, range of motion, functional workspace, goal attainment scale, and surface electromyography.

ELIGIBILITY:
Inclusion Criteria

1. Patients with a confirmed diagnosis of a neuromuscular disease (NMD) by genetic testing, muscle biopsy, or electrodiagnostic studies, presenting with prominent upper limb muscle weakness. Examples include:

   1. Muscular Dystrophies: Duchenne/Becker Muscular Dystrophy (DMD/BMD), Limb-Girdle Muscular Dystrophy (LGMD), Facioscapulohumeral Muscular Dystrophy (FSHD), etc.
   2. Motor Neuron Diseases: Spinal Muscular Atrophy (SMA, Types 2 and 3), Amyotrophic Lateral Sclerosis (ALS, upper limb-dominant), etc.
   3. Peripheral Neuropathies: Charcot-Marie-Tooth (CMT) disease, etc.
   4. Other Neuromuscular Conditions: Including but not limited to cervical spinal cord injury.
2. Aged over 10 years.
3. A score of 2 to 5 on the Brooke Upper Extremity Functional Rating Scale.
4. Manual Muscle Test (MMT) grade of less than 3 for shoulder abduction.
5. Ability to provide written informed consent from the participant and/or their legal representative, indicating willingness to participate in the study.

Exclusion Criteria

1. Unwillingness or inability to provide informed consent.
2. A score of 1 or 6 on the Brooke Upper Extremity Functional Rating Scale.
3. Cognitive impairment severe enough to interfere with the proper use of a shoulder orthosis.
4. Any other condition which, in the opinion of the investigator, would make study participation inappropriate or unsafe for the patient.

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-04-20 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Performance of the upper limb module 2.0 (PUL 2.0) | Before orthosis wear & After orthosis wear and operation
  The Performance of the Upper Limb module (PUL) was specifically designed to assess upper limb function across the spectrum of function in patients with neuromuscular disorder, providing information on three domains of upper limb function (shoulder, middle, distal) and overall upper limb functional abilities. Each domain (shoulder, middle, distal) can be scored separately, and the scores from the three levels are summed up to a maximum of 44 points.
Active Range of motion | Before orthosis wear & After orthosis wear and operation
  Measurement of range of motion is assessed using a goniometer, with the evaluator measuring the active range of motion of the shoulder joint in the same position before and after orthosis wear using the same tool. The measurement is taken with the trunk as the center, and the flexion/extension and abduction/adduction of the humerus are each measured three times, with the average value used.
Functional workspace | Before orthosis wear & After orthosis wear and operation
  Functional workspace analysis consists of 7 movements, where participants are asked to touch specific body parts in sequence: 1. Belly button, 2. Back pocket, 3. Same-side shoulder, 4. Opposite-side shoulder, 5. Mouth, 6. Top of head, 7. Back of head using both right and left hands. Analysis of functional workspace is manually performed based on recordings from 2 video cameras. Scores are assigned on a 4-point scale: 0 indicates inability to perform the task, 1 indicates reaching 0-49% of the target location, 2 indicates reaching 50-99% of the target location, and 3 indicates reaching the target location completely. Cumulative scores are calculated for all movements.
Goal Attainment Scale (GAS) | Before orthosis wear & After orthosis wear and operation
  Setting GAS goals is based on selecting the three most urgent issues among the problems the patient has based on the initial clinical assessment scores, with sufficient consideration given to the opinions of the patient and caregivers through interviews. Subsequently, three specific goals are selected based on the most urgent problems identified by the research team meeting.
Surface electromyography (sEMG) | Before orthosis wear & After orthosis wear and operation
  - Measurement Tasks:
  The following items are selected based on the examiner's judgment, with 3-5 items chosen for measurement:
  i. Shoulder abduction with both arms raised above the head ii. Shoulder height arm raising (based on elbow position) iii. Shoulder flexion at shoulder height iv. Moving wooden blocks v. Pouring water into a cup vi. Placing hand on the abdomen vii. Placing hand in the back pocket viii. Placing hand on the shoulder of the same side ix. Placing hand on the shoulder of the opposite side x. Brushing teeth xi. Brushing front hair
  C. Sensor Attachment Sites:
  - Selected based on the measurement task: i. Anterior/Middle Deltoid (dominant) ii. Biceps Brachii (dominant) iii. Upper Trapezius (dominant) iv. Sternocleidomastoid (dominant) v. External/Internal Oblique Muscles (both sides) vi. Longissimus muscles (both sides)
  D. Sensor Signal Parameters:
  - EMG Parameters: Amplitude after Rectification (RMS), area, percentage ratio of amplitude to RVC during motion.
Heart rate | Baseline and immediately after completing the standard task with the orthosis (approximately 3-4 hour)
  changes in heart rate
Blood pressure | Baseline and immediately after completing the standard task with the orthosis (approximately 3-4 hour)
  changes in blood pressure in systolic and diastolic
Numeral Rating Scale for Pain | Baseline and immediately after completing the standard task with the orthosis (approximately 3-4 hour)
  changes in pain score using Numeral Rating Scale
Box and block test | Baseline and immediately after completing the standard task with the orthosis (approximately 3-4 hour)
  A wooden box with a partition will be used with wooden blocks placed in one side of the box.
  The box is placed longitudinally on a table in front of the participant. The side of the box containing 150 blocks is positioned on the side of the hand being tested.
  The participant is instructed to move as many blocks as possible, one at a time, from the starting compartment to the empty compartment by reaching over the central partition, within a specified time limit.
  The researcher provides a clear demonstration of the task, emphasizing that blocks must clear the partition and enter the opposite side completely.
  A 15-second practice trial is administered first to ensure the participant understands the directions and task demands.
  A 60-second test trial is administered for each hand, starting with the dominant hand. The stopwatch starts when the participant's hand touches the first block and stops precisely at 60 seconds.

CONTACTS AND LOCATIONS:
Overall Officials: Woo Hyung Lee, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, Jongno-gu, South Korea